CLINICAL TRIAL: NCT00340522
Title: Childhood Cancer and Plexiform Neurofibroma Tissue Microarray for Molecular Target Screening and Clinical Drug Development
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904282; 04-C-N282
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-08-11

CONDITIONS: Cancer
Keywords: Sarcoma; Brain Tumor; Embryonal Tumor; Tumor Array; Childhood Cancer; Plexiform Neurofibromas; Drug Screening; Immunohistochemistry
MeSH Terms: conditions — Neoplasms; Sarcoma; Brain Neoplasms; Neoplasms, Germ Cell and Embryonal; Neurofibroma, Plexiform

SUMMARY:
This study will construct tissue microarrays (TMAs) pertaining to childhood cancer. TMA technology is a recently developed one that allows for evaluating hundreds of tissue samples simultaneously on the DNA, RNA, and protein levels. The goal is to identify a potential molecular signature. Cancer drug discovery is currently focused on identifying drugs targeted at the molecular level. Such drugs would be more selective and specific for proteins and signaling pathways that are directly involved in the origin of tumors. However, the origin of cancer among adults differs from that of cancer diagnosed in children. The overall approach by the pharmaceutical industry in developing drugs is not likely to be aimed at low-incidence cancers, such as childhood cancers. Thus, the researchers in this study propose to create a childhood cancer TMA that include specimens from a wide range of solid tumors that present a poor prognosis for patients. This TMA would in turn be used to identify antibodies and lead to developing molecularly targeted drugs that would reach clinical trials in adults.

TMAs are created robotically. Small tissue cores are taken from paraffin-embedded tissue blocks and are implanted into new paraffin blocks. The recipient blocks are then processed to produce several hundred specimens that can be evaluated on a single glass slide. Specimens representing 17 distinct kinds of pediatric solid tumors will be used in this study. Also included will be samples of plexiform neurofibroma-that is, benign growths of nervous and connective tissues.

Tissue specimens will come from patients who were age 25 or younger at the time of diagnosis of their cancer or plexiform neurofibroma. No procedures will be performed for the sole purpose of obtaining tissue for this study.

The TMA developed in this study will not be commercialized. The results for individuals whose tumor specimens are used in the array will not be sent to patients or their treating physicians.

DETAILED DESCRIPTION:
Background: Cancer drug discovery is now focused on identifying molecularly targeted drugs that are more selective and specific for proteins and signaling pathways that are directly involved in tumorigenesis. This new paradigm alters the approach to clinical drug development for childhood cancers because the emphasis is on therapeutic targets present in common epithelially-derived adult cancers, which have a different pathogenesis. The pharmaceutical industry is unlikely to undertake target discovery programs for low incidence cancers, such as childhood cancers. Therefore, a more pragmatic approach to the development of molecularly targeted drugs in children is required.

Objective: Construct a childhood cancer tissue microarrays (TMA) for screening and selecting the most appropriate molecularly targeted agents for clinical development in childhood cancers.

Eligibility: Ten to twenty representative specimens (paraffin blocks) for each of 25 histologically distinct pediatric solid tumors or plexiform neurofibromas will be collected.

Design: Using a robotic arrayer, three 0.6 mm cores from each tissue block will be donated into one of 3 recipient paraffin TMA blocks (CNS tumors, sarcomas, embryonal tumors). Standard immunohistochemical techniques will be applied to 5 micro m sections from the TMA block using validated antibodies directed against specific protein targets of interest. If greater than 8 to 20 tumors from each specific histological type of cancer are positive, there is a 95% probability that the true proportion of positive specimens exceeds 20%. The results of the TMA target assessment will guide in the selection of molecularly targeted drugs for pediatric phase I clinical trials in the POB and Pediatric Phase I/Pilot Consortium and the selection of candidate tumors for activity testing in phase II clinical trials. If clinical responses are observed in phase I or II trials in tumor types that express the target on the TMA, we will return to the original paraffin blocks and perform Laser Capture Microdissection and produce reverse-phase lysate protein microarrays to assess the activation state of targeted signaling pathways and investigate the role of the target protein in tumorigenesis of the responsive childhood cancers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Twenty representative formalin-fixed, paraffin-embedded specimens for each of 17 histologically distinct pediatric solid tumors will be collected from the pathology departments of selected Pediatric Phase I Consortium collaborators.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-09-07; Study Completion 2014-08-11

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C Widemann, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mousses S, Kallioniemi A, Kauraniemi P, Elkahloun A, Kallioniemi OP. Clinical and functional target validation using tissue and cell microarrays. Curr Opin Chem Biol. 2002 Feb;6(1):97-101. doi: 10.1016/s1367-5931(01)00283-6. PMID 11827831
- [Background] Pollock PM, Harper UL, Hansen KS, Yudt LM, Stark M, Robbins CM, Moses TY, Hostetter G, Wagner U, Kakareka J, Salem G, Pohida T, Heenan P, Duray P, Kallioniemi O, Hayward NK, Trent JM, Meltzer PS. High frequency of BRAF mutations in nevi. Nat Genet. 2003 Jan;33(1):19-20. doi: 10.1038/ng1054. Epub 2002 Nov 25. PMID 12447372
- [Background] Weeraratna AT, Becker D, Carr KM, Duray PH, Rosenblatt KP, Yang S, Chen Y, Bittner M, Strausberg RL, Riggins GJ, Wagner U, Kallioniemi OP, Trent JM, Morin PJ, Meltzer PS. Generation and analysis of melanoma SAGE libraries: SAGE advice on the melanoma transcriptome. Oncogene. 2004 Mar 18;23(12):2264-74. doi: 10.1038/sj.onc.1207337. PMID 14755246